CLINICAL TRIAL: NCT06897761
Title: Development of an Interactive Digital Respiratory Game and Device and Investigation of Its Effectiveness in Children With Bronchiectasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Hilal Denizoğlu Külli, Assoc. Prof., Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hilal Denizoglu Kulli
Record Dates: First submitted 2024-09-18; First posted 2025-03-27 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Bronchiectasis
Keywords: respiratory game, Active Cycle of Breathing Techniques; bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Game Group (Experimental): The participants will perform the interactive digital game.
  Interventions: Device: Interactive Digital Respiratory Game; Other: home-based exercise training
- Control Group (Active Comparator): The participants will perform home based exercise
  Interventions: Other: home-based exercise training

INTERVENTIONS:
Device: Interactive Digital Respiratory Game — With the development of technology and digitalization, Digital Respiratory Games (DRG) offer an alternative solution. DRGs, with their difficulty levels, provide a platform for progression, offering a fun and engaging experience that enhances patient adherence to therapy through storytelling and user interaction. The absence of a locally made DRG in Turkey, despite the chronic respiratory diseases impact, has led to the need for an interactive DRG with personalized features. The developed interactive DRG and device will be Turkey first interactive DRG example, designed to respond to different respiratory maneuvers. The developed DRG and device will detect the lung volume and flow rates and allow for the real-time execution of maneuvers within the Active Cycle of Breathing Techniques (ACBT) in a playful environment.
  Arms: Breathing Game Group
Other: home-based exercise training — Patients in the home-based exercise training group will be asked to perform the active breathing techniques cycle, which is an airway clearance technique, twice a day, 7 days a week, for 20 minutes each, for 8 weeks and to follow the program that includes physical activity recommendations. Patients who use mucolytic and/or nebulized drugs such as hypertonic saline or mannitol will be instructed to perform nebulization before performing the active breathing techniques cycle.
  Other Names: chest physiotherapy

SUMMARY:
Our study aims to develop a personalized interactive digital breathing game and device that can be produced in our country and to provide daily airway cleaning treatment at home via mobile phone or computer without the need for a physiotherapist or healthcare professional with the use of an interactive digital breathing game.

DETAILED DESCRIPTION:
The disruption of airway clearance may lead to obstruction, respiratory infections, gas exchange deterioration, and an increase in mortality and morbidity. Airway clearance is especially crucial in children with bronchiectasis. Postural drainage, manual techniques, positive expiratory pressure, and chest oscillation devices are among airway clearance techniques. The repetitive and frequent use of these techniques strengthens adherence to therapy. With the development of technology and digitalization, Digital Respiratory Games (DRG) offer an alternative solution. DRGs, with their difficulty levels, provide a platform for progression, offering a fun and engaging experience that enhances patient adherence to therapy through storytelling and user interaction. The absence of a locally made DRG in Turkey, despite the chronic respiratory diseases impact, has led to the need for an interactive DRG with personalized features. The developed interactive DRG and device will be Turkey first interactive DRG example, designed to respond to different respiratory maneuvers. The developed DRG and device will detect the lung volume and flow rates and allow for the real-time execution of maneuvers within the Active Cycle of Breathing Techniques (ACBT) in a playful environment. The interactive DRG will enable airway clearance at home and in daily life, without the need for a physiotherapist, in a progressive, fun, and environmentally compatible manner, adjusted to capacity of the user. The interactive DRG and device possess useful model or patentable value and unique features. The aim of the study is to investigate the effectiveness of the locally produced interactive DRG and device in children with bronchiectasis.

The accepted and supported 2022-B-03 call for TUSEB project includes producing personalized interactive digital respiratory games and examining their effects in children with bronchiectasis. A total of 40 children (n=20 in the DRG group and n=20 in the control group) will participate in the study. Participants will perform physical activity exercises specific to their group's treatment protocol, twice a day for 7 days a week, over 8 weeks. Following treatment, their lung function, peripheral respiratory muscles, capacity, treatment adherence, quality of life, and treatment satisfaction will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 7-18 years
* Clinically stable
* No exacerbations or infections
* Possesses a computer, tablet, or mobile phone

Exclusion Criteria:

* Participation in a supervised physiotherapy and rehabilitation program within the last 6 months
* History of lung or liver transplant
* Presence of any cognitive impairment that would hinder the use of the system
* Changes in medical treatment during the study
* Presence of concurrent cardiac, orthopedic, or neurological diseases

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2025-12-07 (Actual); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Test | baseline and within 1 week after intervention
  6MWT is defined as a submaximal test that can be easily applied in healthy or unhealthy individuals and is evaluated as an indicator of exercise capacity and walking capacity as well as many cardiovascular diseases. The 6MWT is referred to as the "Gold Standard" test of walking capacity. The aim of this test is to reach the longest possible walking distance at the end of six minutes. The standard protocol is applied in a 30-meter uninterrupted corridor or open area. It is recommended to repeat the 6MWT three times on the same day with a one-hour rest interval; the maximum walking distance is taken into account.
Evaluation of Expiratory Muscle Strength | baseline and within 1 week after intervention
  Inspiratory and expiratory respiratory muscle strength will be evaluated by measuring maximal mouth pressure. Maximal mouth pressure will be measured using the Micro RPM brand (Micro Medical; England) portable electronic mouth pressure measurement device, in accordance with ATS/ERS criteria. Maximal expiratory pressure (MEP) will be measured to assess expiratory muscle strength.
Evaluation of Inspiratory Muscle Strength | baseline and within 1 week after intervention
  Inspiratory and expiratory respiratory muscle strength will be evaluated by measuring maximal mouth pressure. Maximal mouth pressure will be measured using the Micro RPM brand (Micro Medical; England) portable electronic mouth pressure measurement device, in accordance with ATS/ERS criteria. Maximal inspiratory pressure (MIP) will be measured to assess inspiratory muscle strength,.

SECONDARY OUTCOMES:
Evaluation of Quality of Life | baseline and within 1 week after intervention
  The general quality of life questionnaire selected for children is the PedsQoL - Pediatric Quality of Life Inventory (PQLI).
  This scale consists of 23 items and 4 subscales, including 8 items measuring physical functioning, 5 items measuring emotional functioning, 5 items measuring social functioning and 5 items assessing school functioning. The minimum and maximum scores of the scale are 0 and 100. Higher scores present better quality of life.
Evaluation of Cough | baseline and within 1 week after intervention
  The Leicester Cough Questionnaire (LCQ) consists of 19 questions under 3 subdomains (physical, psychological, and social), is a quality of life questionnaire related to chronic cough and health. It is rated on a 7-point Likert scale. Higher scores show better condition.
Assessment of Sleep Quality | baseline and within 1 week after intervention
  In our project, sleep quality will be assessed with the "Pediatric Sleep Scale" developed by Chervin et al. and Turkish validation and reliability by Yüksel et al. This scale, completed by parents, contains information about 22 sleep-related symptoms. Each positive symptom is given a score of "1" and a score of 8 or more on the scale is considered as "sleep disordered sleep".
Evaluation of Peripheral Muscle Strength | baseline and within 1 week after intervention
  Quadriceps muscle strength will be evaluated to assess peripheral muscle strength. Muscle strength will be measured using the MicroFET®; brand (Hoggan Scientific; USA) electronic handheld dynamometer. Each muscle strength assessment will be performed with the participant in a seated position with back support, following standard test procedures. The muscle strength test will be repeated three times for the participant's dominant extremity, and the average of the measurements will be recorded.
Respiratory Function Test- FEV1 value | baseline and within 1 week after intervention
  Pulmonary function will be evaluated with a spirometer according to the American Thoracic Society and European Respiratory Society criteria. The device replaces the hand-held flow sensor, traditionally placed in the mouth, with the same sensor being secured to the face using straps and a mask. Participants will be asked to take a deep breath and then perform a strong and complete exhalation. This maneuver will be repeated three times, and the best of the three measurements, with a difference of less than 0.150 L between them, will be recorded. Forced expiratory volume in 1 second (FEV1) will be recorded. When data such as age, gender, race, height, and weight are entered into the device, the expected values of all parameters will be calculated based on normative values.
Respiratory Function Test- FVC value | baseline and within 1 week after intervention
  Pulmonary function will be evaluated with a spirometer according to the American Thoracic Society and European Respiratory Society criteria. The device replaces the hand-held flow sensor, traditionally placed in the mouth, with the same sensor being secured to the face using straps and a mask. Participants will be asked to take a deep breath and then perform a strong and complete exhalation. This maneuver will be repeated three times, and the best of the three measurements, with a difference of less than 0.150 L between them, will be recorded. Forced vital capacity (FVC) will be recorded. When data such as age, gender, race, height, and weight are entered into the device, the expected values of all parameters will be calculated based on normative values.
Respiratory Function Test- FEV1/FVC | baseline and within 1 week after intervention
  Pulmonary function will be evaluated with a spirometer according to the American Thoracic Society and European Respiratory Society criteria. The device replaces the hand-held flow sensor, traditionally placed in the mouth, with the same sensor being secured to the face using straps and a mask. Participants will be asked to take a deep breath and then perform a strong and complete exhalation. This maneuver will be repeated three times, and the best of the three measurements, with a difference of less than 0.150 L between them, will be recorded. Tiffeneau ratio (FEV1/FVC) will be recorded.
Respiratory Function Test- PEF value | baseline and within 1 week after intervention
  Pulmonary function will be evaluated with a spirometer according to the American Thoracic Society and European Respiratory Society criteria. The device replaces the hand-held flow sensor, traditionally placed in the mouth, with the same sensor being secured to the face using straps and a mask. Participants will be asked to take a deep breath and then perform a strong and complete exhalation. This maneuver will be repeated three times, and the best of the three measurements, with a difference of less than 0.150 L between them, will be recorded. Peak expiratory flow (PEF),will be recorded. When data such as age, gender, race, height, and weight are entered into the device, the expected values of all parameters will be calculated based on normative values.

OTHER OUTCOMES:
Evaluation of Participation in the Program | baseline and within 1 week after intervention
  Participation in the 8-week program will be monitored with an exercise diary that will be given to the patients. The diary will include information on whether the patient completed the program completely and the duration, number and frequency of the exercises.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided